CLINICAL TRIAL: NCT06429670
Title: Real World Use of Azacitidine and Venetoclax in Acute Myeloid Leukemia in Frontline and Relapse/Refractory Settings: a Multicentric Study From French AURAML Group
Brief Title: Real World Use of Azacitidine and Venetoclax in Acute Myeloid Leukemia in Frontline and Relapse/Refractory
Acronym: VENAURA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0521
Record Dates: First submitted 2024-05-13; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; azacitdine; venetoclax; MRD
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Azacytidine and venetoclax treated patients: Adult patients with acute myeloid leukemia treated by AZACYTIDINE and VENETOCLAX in frontline and relapse/refractory settings

SUMMARY:
Azacytidine and venetoclax combination regimen (AZA/VEN) is the standard of care in frontline acute myeloid leukemia (AML) settings for unfit to intensive chemotherapy patients. AZA/VEN combination regiment was approved in France in 2021 but was already used in outlabel fashion since 2019. However, AZA/VEN is also associated with an increased hematological toxicity compared to azacytidine alone. In this context, alternative AZA/VEN regimens emerged progressively based on each physician experience and local procedures. Moreover, AZA/VEN is also recognized as a valuable therapeutic option in relapse/refractory settings. In this multicentric study, the investigators aimed to evaluate the efficacy and safety of various AZA/VEN regimen in frontline and relapse/refractory (R/R) patients diagnosed with AML in real life setting.

The investigators will retrospectively analyze clinical outcome of patients from 11 different French centers (Saint-Etienne, Clermont-Ferrand, Lyon (Hopital Lyon Sud, Centre Léon Bérard), Vichy, Annecy, Chambery, Valence, Bourgoin-Jallieu, Grenoble, Roanne) in Auvergne Rhône Alpes (AURA) region, between January 2019 and December 2023. Composite complete remission was defined as in VIALE-A trial. Measurable residual disease (MRD) negativity was defined as ≤ 10-3 by flow cytometry (on bone marrow) and/or ≤ 10-4 for NPM1 by RT-qPCR.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Acute myeloid leukemia patients at diagnostic, in relapse/refractory settings, or MRD relapse.
* receiving AZA/VEN combination regimen

Exclusion Criteria:

* Another VEN combination chemotherapy
* AZA/VEN initiation prior January 2019 and after December 2023
* Opposition to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every adult patients ( >18 years old) with a diagnostic of AML treated by the association of AZACYTIDINE and VENETOCLAX between January 2019 and December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | up to 5 months
  Overall survival corresponds to time to death from the initiaiton of AZA/VEN, regardless of disease recurrence.

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Centre Hospitalier Pierre Oudot | Groupement hospitalier Nord, Bourgoin
  - METROPOLE SAVOIE - SITE CHAMBERY, place Lucien Biset,, Chambéry
  - CHU Clermont-Ferrand Site Estaing, Clermont-Ferrand
  - Centre Hospitalier Annecy Genevois, Épagny
  - CHU Grenoble Alpes, La Tronche
  - Centre Léon Bérard, Lyon
  - Hospices Civils de Lyon, Lyon
  - Centre Hospitalier de Roanne, Roanne
  - CHU de Saint-Étienne Hôpital Nord, Saint-Priest-en-Jarez
  - Centre Hospitalier de Valence, Valence
  - Ch de Valence, Valence
  - Hopital Vichy, Vichy

IPD SHARING:
Plan to Share IPD: No